CLINICAL TRIAL: NCT05360810
Title: Comparison of Wei Nasal Jet Tube vs Gastro Laryngeal Tube in Endoscopic Retrograde Cholangiopancreatography: A Prospective, Randomized, Observational Study
Brief Title: Wei Nasal Jet Tube vs Gastro Laryngeal Tube in Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Harun UYSAL, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: BezmialemVakifU
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Supraglottic Airway Efficiency; Airway Complication of Anesthesia; Airway Aspiration; Complication of Anesthesia; Esophagus Injury; Endoscopic Ergonomics; ERCP Airway Management; Bleeding Nose; Bronchospasm
Keywords: Wei Nasal Jet Tube; Gastro-laryngeal tube; ERCP; Airway Complication; Hipoxia
MeSH Terms: conditions — Epistaxis; Bronchial Spasm

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) closed envelope technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wei Nasal Jet Tube Group (Group W) (Active Comparator): After induction of anesthesia, the Wei Nasal Jet Tube was placed in the patients.
  Interventions: Device: Wei Nasal Jet Tube
- Gastro-Laryngeal Tube Group (Group G) (Active Comparator): After the induction of anesthesia, the Gastro Laryngeal Tube was placed in the patients.
  Interventions: Device: Gastro Laryngeal Tube

INTERVENTIONS:
Device: Wei Nasal Jet Tube — comparing efficiency and complications of second generation airway devices which can use for gastrointestinally procedures
  airway devices which can use for gastrointestinal procedures
  Other Names: Comparison of LMA Gastro Airway® and Gastro-Laryngeal Tube in patients who will ERCP procedures.
  Arms: Wei Nasal Jet Tube Group (Group W)
Device: Gastro Laryngeal Tube — comparing efficiency and complications of second generation airway devices which can use for gastrointestinally procedures
  Other Names: Comparison of LMA Gastro Airway® and Gastro-Laryngeal Tube in patients who will ERCP procedures.
  Arms: Gastro-Laryngeal Tube Group (Group G)

SUMMARY:
The most common adverse event in endoscopic procedures is hypoxia. Different airway devices have been investigated in the literature to prevent hypoxia. This study aimed to compare the efficacy and procedural performance of two different airway (GLT and WNJ) devices in ERCP procedures.

DETAILED DESCRIPTION:
ERCP is a procedure that requires intolerable positioning, prolonged air insufflation, and deep levels of anesthesia. The procedure can be performed under general anesthesia or with deep sedation. It becomes more difficult to maintain airway patency in the prone position under deep sedation. Clinicians prefer supraglottic airway devices developed for endoscopic procedures. GLT requires a deeper level of anesthesia. WNJ, on the other hand, can be tolerated with less depth levels of anesthesia. It has been reported in the literature that GLT and WNJ are effective in maintaining patent airway and preventing hypoxia in ERCP procedures. However, both airway devices have not been compared for airway efficiency and ERCP procedure condition.

In this study, the investigators aimed to compare airway efficiency and procedure condition using GLT and WNJ.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1-2
* Elective Procedures
* Body mass index 18.5 - 35 kg/m2

Exclusion Criteria:

* High risk of pulmonary aspiration
* Pregnancy
* Anesthesic drug allergies
* Difficult airway or facial deformities
* Height <155 cm
* Alcohol or narcotic drug usage
* Restrictive or obstructive pulmonary diseases
* Hepatic cardiac or renal failure
* Neurologic or cognitive deficiencies.
* Previous cervical surgery or cervical radiotherapy
* Previous esophagus surgery
* Psychotic problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Hypoxia İncidence | Intra-operative; after device insertion
  Hypoxia is defined as SpO2 <92% at any time.
Endoscopist Satisfaction Analysis: Score | Intra-operative, during the procedure
  It is determined by the endoscopist according to the endoscopy satisfaction scale according to the maneuverability of the duodenoscope and the number of insertion attempts. (0-10 Points) The endocopist satisfaction score is scored on a minimum score of 0 and a maximum of 10 points. A score of 0 means I am not satisfied at all, a score of 10 means very satisfied. A higher score indicates higher satisfaction.

SECONDARY OUTCOMES:
Blood staining on the device | Immediately after removing the supraglottic airway device
  Whether there is blood on the supraglottic airway device or not
Presence of sore throat | One hour after extubation
  Sore throat if present, was classified as mild, moderate or severe.
Incidence of hypercapnia | Intra-operative; after device insertion
  Hypercapnia is EtCO2 >45 mmHg at any time during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Harun Uysal, M.D., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)